CLINICAL TRIAL: NCT05084105
Title: Cannabis Use and Risk of Falling in Older Adults: an Observation Study
Brief Title: Cannabis and Aging
Status: Completed | Type: Observational
Sponsor: Thorsten Rudroff (Other)
Responsible Party: Sponsor-Investigator, Thorsten Rudroff, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201909808
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Cannabis Use
Keywords: Cannabis; Aging; Falls; Brain Glucose Uptake
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cannabis Group: A total of 30 older (age 50-80 years) men and women who are using cannabis.
- Control Group: A total of 30 older (age 50-80 years) men and women who are not using cannabis.

SUMMARY:
With increased availability and use of cannabis by older adults aged ≥ 50 years, a rigorous evaluation of the benefits and risks of cannabis use in these individuals is necessary. Our proposed project will investigate whether older adults who initiate cannabis use after the age of 50 are at an increased risk of fall and what are the underlying mechanisms. We will measure motor and cognitive function in older cannabis users and nonusers and we will use positron emission tomography to determine brain activity and how it is associated with fall risk.

DETAILED DESCRIPTION:
The prevalence of cannabis use has increased significantly in recent years among US adults aged 50 years and older. With increased availability and use of cannabis by older adults, a rigorous evaluation of the benefits and risks of cannabis use in these individuals is necessary. Aging is characterized by physiological and social changes that make older adults vulnerable to chronic disease and geriatric conditions, including cognitive impairment and falls. Unintentional falls are a common event for older adults and a major cause of morbidity and mortality linked with a decline in functional status and disability. Moreover, falls and cognitive impairment are a "well-known couple"; as older adults with moderate to severe cognitive impairment have a higher risk of falls, with an annual incidence of around 60-80%, which is twice the rate of cognitively normal older adults. Impaired cognitive function is an effect of cannabis use, and there is increasing evidence that those effects may persist later in life. Therefore, the physiological effects of chronic cannabis use may further increase falls in older adults via alterations in gait and cognition. Studies have shown reduced neural activity in the frontal brain networks and associations with increased fear of falling in older adults. It is also known that in regular cannabis users, the effects of cannabis may have an impact on cognitive-motor skills and brain mechanisms that modulate coordinated movement. The goal of this application is to investigate the neural correlates of fall risk and cognitive and motor function in individuals who initiate drug use after the age of 50. We will use FDG-PET to determine brain activity. Fall risk and cognitive/motor function will be assessed with the measures from the NIH Toolbox and a fall risk model. Our central hypothesis is that older chronic cannabis users are at a higher fall risk than older non-users, which is associated with reduced cerebral FDG uptake. These results are expected to provide critical and timely data to the public and health professionals regarding the effects of self-directed cannabis use on increased fall risk and if clinicians need to assess cannabis use when determining fall risk and deciding prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* 50-80 years
* Healthy enough to complete the protocol based on information obtained from a clinical exam and past medical history, such as cardiovascular diseases.
* Comprehension of the protocol as indicated by an ability to respond to questions about the study after reading the consent form.
* Able to use and be contacted by telephone.
* Able to speak, read, and understand English, and complete a questionnaire in English

Exclusion Criteria:

* Presence of pacemakers, aneurysm clips, artificial heart valves, metallic prostheses
* Pregnancy
* History of significant traumatic brain injury
* Unable to lie flat for the study imaging

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 30 older (age 50-80 years) men and women who are using cannabis and 30 controls who are non-users, will be recruited.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Fall Risk | Through study completion, on average 1 year
  The following equation for the prediction of falls will be used:
  Likelihood of falling (%) = (exp (-7.519 + 0.026(reaction time) - 0.071(ABC1) - 2.139(Berg 14))) / (1 + exp (-7.519 + 0.026(reaction time) - 0.071(ABC1) - 2.139(Berg 14)) ×100)
Brain activity PET Imaging | Through study completion, on average 1 year
  To investigate cerebral glucose uptake in older chronic cannabis users and non-users

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Health and Human Physiology, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No